CLINICAL TRIAL: NCT03842371
Title: Metabolism of Branched-chain Amino Acids in Monocyte and Macrophage During Sepsis
Brief Title: Metabolism of Branched-chain Amino Acids in Monocyte/Macrophage During Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Clinical Professor, West China Hospital
Other Study IDs: 2018-081
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Sepsis Syndrome
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sepsis with type 2 diabetes: Sepsis patients with type 2 diabetes
  Interventions: Other: Metabolic level of BCAAs in monocytes and macrophages
- Sepsis without type 2 diabetes: Sepsis patients without type 2 diabetes
  Interventions: Other: Metabolic level of BCAAs in monocytes and macrophages
- Volunteers: Healthy volunteers
  Interventions: Other: Metabolic level of BCAAs in monocytes and macrophages

INTERVENTIONS:
Other: Metabolic level of BCAAs in monocytes and macrophages — Metabolic level of BCAAs in monocytes and macrophages

SUMMARY:
The current project was designed to examine the metabolic level of branched-chain amino acids in plasm and monocyte/macrophage, and its role in immune dysfunction during sepsis.

DETAILED DESCRIPTION:
In this study, the investigators will collect the peripheral blood of 1,3,7,14 day after diagnose of sepsis. Then, the concentration of branched-chain amino acids(BCAAs) in monocytes and plasma, and the expression of BCAAs metabolic enzymes in monocytes will be determined. Additionally, the inflammatory cytokines, e.g., Interleukin-1β (IL-1β), Tumor necrosis factor-α (TNF-α), Interleukin-10 (IL-10）, the chemokines macrophage inflammatory proteins 1α and 1β (MIP-1α and 1β) in the peripheral blood and the phagocytic function of monocytes will also be detected. The current project was designed to examine the metabolic level of branched-chain amino acids in plasm and monocyte/macrophage, and its role in immune dysfunction during sepsis.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with sepsis, with or without type 2 diabetes
* healthy volunteers

Exclusion Criteria:

* patients with immunodeficient diseases
* patients who accept glucocorticoid or immunosuppressant
* patients with an age younger than 18 years
* patients who cannot provide the informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed as sepsis, with or without type 2 diabetes.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-02-11 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Intracellular levels of branched-chain amino acids in monocytes | up to 14 day after diagnose of sepsis
  BCAAs Assay Kit will be used to measure the intracellular levels of BCAAs in monocytes.

SECONDARY OUTCOMES:
Plasma levels of branched-chain amino acids | 1,3,5,7,10,14 day after diagnose of sepsis
  BCAAs Assay Kit will be used to measure the plasma levels of BCAAs.
The expression of branched-chain amino acid aminotransferase in monocytes | 1,3,5,7,10,14 day after diagnose of sepsis
  The expression of branched-chain amino acid aminotransferase in monocytes will be determined by qPCR and western blot.
The expression of branched-chain α-ketoacid dehydrogenase in monocytes | 1,3,5,7,10,14 day after diagnose of sepsis
  The expression of branched-chain α-ketoacid dehydrogenase in monocytes will be determined by qPCR and western blot.
The expression of PP2Cm in monocytes | 1,3,5,7,10,14 day after diagnose of sepsis
  The expression of mitochondrial-targeted phosphatase, PP2Cm in monocytes will be determined by qPCR and western blot.
The plasma level of IL-1β | 1,3,5,7,10,14 day after diagnose of sepsis.
  The plasma level of IL-1β will be determined by ELISA kit.
The plasma level of TNF-α | 1,3,5,7,10,14 day after diagnose of sepsis.
  The plasma level of TNF-α will be determined by ELISA kit.
The plasma level of IL-10 | 1,3,5,7,10,14 day after diagnose of sepsis.
  The level of IL-10 will be determined by ELISA kit.
The plasma level of chemokine MIP-1α. | 1,3,5,7,10,14 day after diagnose of sepsis.
  The plasma level of chemokine MIP-1α will be determined by ELISA kit.
The plasma level of chemokine MIP-1β. | 1,3,5,7,10,14 day after diagnose of sepsis.
  The plasma level of chemokine MIP-1β will be determined by ELISA kit.
The phagocytic index of monocytes. | 1,3,5,7,10,14 day after diagnose of sepsis.
  The phagocytic index of monocytes will be determined by a E.coli Phagocytosis Assay Kit.

IPD SHARING:
Plan to Share IPD: No